CLINICAL TRIAL: NCT04137640
Title: Palbociclib + Letrozole Versus Epirubicin + Cyclophosphamide and Sequential Docetaxel as Neoadjuvant Chemotherapy for Postmenopausal Estrogen Receptor-positive Breast Cancer: a Prospective Randomized Controlled Double-blind Phase IV Trial
Brief Title: Palbociclib + Letrozole Versus Epirubicin + Cyclophosphamide and Sequential Docetaxel as Neoadjuvant Chemotherapy
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Caigang Liu, Principal Investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Shengjing-LCG003
Record Dates: First submitted 2019-10-22; First posted 2019-10-24 (Actual); Last update posted 2021-07-20 (Actual); Status verified 2021-07

CONDITIONS: Breast Cancer
Keywords: adjuvant chemotherapy; estrogen receptor; palbociclib; letrozole
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Cyclophosphamide

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- endocrine group (Other): 76 postmenopausal estrogen receptor-positive LABC patients with low Ki67 expression will beassigned into endocrine group.
  Interventions: Drug: palbociclib combined with letrozole
- chemotherapy group (Other): 76 postmenopausal estrogen receptor-positive LABC patients with low Ki67 expression will beassigned into chemotherapy group
  Interventions: Drug: epirubicin combined with cyclophosphamide and sequential docetaxel

INTERVENTIONS:
Drug: palbociclib combined with letrozole — Endocrine group will receive palbociclib combined with letrozole: palbociclib (Pfizer Manufacturing Deutschland GmbH, Freiburg, Germany; license number: H20180040) 125 mg/d, every 28 days as a cycle (medication for 3 consecutive weeks and withdrawal for 1 week); letrozole (Novartis Pharma Schweiz AG, Stein, Switzerland; license number: H20140149) 2.5 mg/d, for 6 consecutive months.
  Other Names: Endocrine group
  Arms: endocrine group
Drug: epirubicin combined with cyclophosphamide and sequential docetaxel — Chemotherapy group will receive epirubicin combined with cyclophosphamide and sequential docetaxel: epirubicin (Pfizer Wuxi Pharmaceutical Plant, Wuxi, China; license number: GYZZ H20000496), 90 mg/m2, intravenously, for 120 minutes, once every four weeks, totally four times; cyclophosphamide (Baxter Oncology GmbH, Halle, Germany; license number: H20160468), 600 mg/m2, once every four weeks, totally four times; sequential docetaxel (Sanofi-aventis Deutschland GmbH, Frankfurt am Main, Germany; license number: GYZZ J20150083) 75 mg/m2, intravenously, for 120 minutes, once every four weeks, totally four times.
  Other Names: Chemotherapy group
  Arms: chemotherapy group

SUMMARY:
With the development of neoadjuvant therapy for tumors, neoadjuvant chemotherapy (NAC) has become one of the most common and effective methods for preoperative systemic treatment of locally advanced breast cancer (LABC). Although epirubicin combined with cyclophosphamide and sequential docetaxel has been widely recognized as the first-line NAC for LABC, there are still some inoperable LABCs that are insensitive to chemotherapy and miss the opportunity of surgery, especially those with luminal A and low expression of Ki67. Therefore, neoadjuvant endocrine therapy has important clinical value for such patients. At present, the combination of aromatase inhibitor drugs and cyclin dependent kinase 4/6 can significantly improve the prognosis and survival of LABC compared with aromatase inhibitor monotherapy. However, whether inoperable LABC patients, especially those who are not susceptible to chemotherapy, can choose the combination of aromatase inhibitor drugs and cyclin dependent kinase 4/6 as neoadjuvant endocrine therapy to replace NAC remains unclear. Because the main principle of endocrine therapy is to induce tumor cell cycle arrest, leading to apoptosis of tumor cells, the effect is slower than that of chemotherapy. In addition, whether endocrine therapy can replace chemotherapy as a new adjuvant treatment for patients with inoperable LABC to improve the operability rate has not yet been fully evidenced. Therefore, this trial aims to conduct the prospective randomized controlled phase IV clinical trial of palbociclib combined with letrozole versus epirubicin combined with cyclophosphamide and sequential docetaxel as NAC to prove the efficacy of palbociclib combined with letrozole in postmenopausal estrogen receptor-positive LABC patients with low Ki67 expression.

DETAILED DESCRIPTION:
reast cancer is one of the most prevalent malignant tumors in women, accounting for 23% of all malignant tumors. Approximately 1.3 million people are diagnosed with breast cancer every year in the world, and approximately 400,000 people die of breast cancer. The overall median survival time of patients with advanced breast cancer is only 2-3 years, and the 5-year survival rate is only about 20%. At present, a considerable number of patients are diagnosed as LABC at the time of initial diagnosis. Because of the wide range of lesions or poor lymph node status, surgical treatment is very difficult, and even some patients cannot be operated on.

With the development of neoadjuvant therapy for tumors, NAC has become one of the most common and effective methods for preoperative systemic treatment of LABC. The 2018 V2 version of the National Comprehensive Cancer Network guidelines for breast cancer diagnosis clearly states that preoperative chemotherapy for LABC should be based on an anthracyclines and can be combined with taxanes, but about 20% of LABC patients are not sensitive to this protocol. Heller et al. performed NAC with 5-fluorouracil + epirubicin + cyclophosphamide for 6 weeks in 88 patients with LABC, and the total effective rate was 78%. After 4 weeks of docetaxel treatment in patients with poor response, approximately 10% of patients are still not sensitive. In addition, many studies in and outside China have pointed out that the NAC effect in some estrogen receptor-positive LABC patients, especially postmenopausal luminal A patients, is worse than that of estrogen receptor negative or Ki67 overexpression patients. Ring et al. treated 435 cases of breast cancer with NAC of doxorubicin/cyclophosphamide or cyclophosphamide/methotrexate/fluorouracil. Pathological complete remission rate was 8.1% in estrogen receptor-positive patients and 21.6% in estrogen receptor negative patients. Similar results were obtained in NSABP B-27 test, with the ratio of 8.3% and 16.7% respectively. Simultaneously, Fashing et al. found that the pathological complete remission of patients with relatively high Ki67 after NAC with anthracyclines combined with taxanes was higher than that of patients with low Ki67. Many clinical studies in China have also obtained similar results; that is, the low expression of Ki67 indicates that the effect of NAC in LABC is not good.

Considering the above situation, some scholars gradually introduce endocrine therapy into the NAC of postmenopausal estrogen receptor-positive LABC, namely neoadjuvant endocrine therapy. At present, neoadjuvant endocrine therapy is practical and feasible for breast cancer with large tumors and positive hormone receptor. Simultaneously, the efficacy of the third-generation aromatase inhibitors is better than that of tamoxifen. Z1031 clinical trial of 381 patients with stage II or III postmenopausal estrogen receptor-positive breast cancer in the United States preliminarily confirmed that the third-generation aromatase inhibitors are currently the first choice of effective neoadjuvant endocrine therapy for postmenopausal estrogen receptor-positive breast cancer. However, 30% to 40% of breast cancer patients receiving endocrine therapy still have disease progression due to drug resistance, which is very disadvantageous for LABC patients. The emergence of cyclin dependent kinase 4/6 inhibitors has given hope to such patients. In the guidelines for advanced breast cancer, Cardoso et al. suggested that a first-line treatment with aromatase inhibitors combined with cyclin dependent kinase 4/6 inhibitors should be preferred. In a phase II randomized controlled trial to explore the treatment of estrogen receptor-positive and epidermal growth factor receptor-2-negative advanced breast cancer by combination of palbociclib, a cyclin dependent kinase 4/6 inhibitor, and letrozole, an aromatase inhibitor, the results found that the former could significantly prolong progression-free survival of hormone receptor-positive advanced breast cancer. Therefore, in February 2015, the US Food and Drug Administration approved the combination of palbociclib and letrozole for first-line treatment of hormone receptor-positive advanced breast cancer. However, for inoperable LABC patients, especially those who are not sensitive to chemotherapy, whether the combination of palbociclib and letrozole can be used as a neoadjuvant endocrine therapy instead of NAC is not clear. Although there are relatively few controlled studies on neoadjuvant endocrine therapy and NAC, the existing evidence suggests that the high level of Ki67 in hormone receptor-positive cases indicates that the effect of chemotherapy is better than that of endocrine therapy, but the adverse reaction rate of chemotherapy is high, especially for LABC or older and infirm patients, while neoadjuvant endocrine therapy can achieve similar effect to NAC. Therefore, the efficacy of palbociclib combined with letrozole as neoadjuvant endocrine therapy is still worth looking forward to. Because the principle of endocrine therapy is mainly to induce tumor cell cycle arrest, leading to apoptosis of cancer cells, so the effect is slower than that of chemotherapy. In addition, whether the efficacy can replace chemotherapy as NAC in inoperable LABC patients to improve the operability rate has not yet been fully evidenced.

Therefore, this trial aims to conduct the prospective randomized controlled phase IV clinical trial using palbociclib combined with letrozole versus epirubicin combined with cyclophosphamide and sequential docetaxel as NAC to prove the efficacy of palbociclib combined with letrozole in postmenopausal estrogen receptor-positive LABC patients with low Ki67 expression.

ELIGIBILITY:
Inclusion Criteria:

* pathological examination confirms estrogen receptor positive, and Ki67 < 30% in breast cancer patients;
* postmenopausal women;
* tumor size stage ≥ T3, or lymph node stage ≥ N2, or ipsilateral upper extremity edema or the extent of lesions exceeds the scope of radical surgery;
* Karnofsky functional status score ≥ 70;
* normal findings of blood examination, normal liver and kidney functions, and basically normal electrocardiogram results before chemotherapy;
* age range from 18-70 years old.

Exclusion Criteria:

* history of anti-tumor treatment;
* inflammatory breast cancer or occult breast cancer;
* stage IV breast cancer;
* history of other malignant tumors;
* severe vital organ dysfunction, such as heart, liver and kidney or poor constitution cannot tolerate chemotherapy, or the treatment plan change due to intolerance during chemotherapy;
* cannot comply with the treatment because of mental and neurological diseases;
* dexamethasone contraindications or severe allergies to any drug in NAC;
* receiving NAC, but it is judged to be ineffective after two cycles of treatment, and other programs are forced to be used or chemotherapy is stopped to receive surgery;
* participation in other clinical trials.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 152 (Estimated)
Dates: Start 2021-07-19 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Clinical Response | 5 years after treatment
  Clinical response will be evaluated 5 years after treatment according to the regression of tumors. Tumor regression will be assessed according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1).

SECONDARY OUTCOMES:
Breast-conserving rate | 6 months after treatment
  The percentage of patients receiving breast-conserving surgery 6 months after treatment
Operable rate | 6 months after treatment
  The percentage of patients who can undergo surgery 6 months after treatment
Ki67 expression in tumor tissues | Before treatment and 6 months and 5 years after treatment
  Immunohistochemical staining will be used before treatment and 6 months and 5 years after treatment
Miller-Payne grading system | Before treatment, 6 months and 5 years after treatment
  Assessment will be conducted before treatment, 6 months and 5 years after treatment. Grade 1: no reduction in the overall cellularity; grade 2: a minor loss of tumor cells but overall cellularity still high; up to 30% loss; grade 3: between an estimated 30% to 90% reduction in tumor cells; grade 4: more than 90% loss of tumor cells; grade 5: no malignant cells identifiable in sections from the site of tumor; however, ductal carcinoma in situ may be present.
Preoperative endocrine prognostic index | 6 months and 5 years after treatment
  Assessment will be conducted 6 months and 5 years after treatment. Preoperative endocrine prognostic index is an independent predictor for breast cancer recurrence, based on tumor size, lymph node status, estrogen receptor status and Ki67 positive rate. The total score is 12. The higher the score, the worse the prognosis is.
Progression-free survival | Within 5 years of follow-up
  Progression-free survival refers to the time from random assignment in a clinical trial to disease progression or death from any cause
Overall survival | Within 5 years of follow-up
  Overall survival refers to the time from group assignment to death
Adverse events | in 5 years
  Any untoward medical occurrence in a patient and which does not necessarily have a causal relationship with this treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Caigang Liu, M.D., Ph.D., Principal Investigator — Shengjing Hospital
Locations (1):
- Shengjing Hospital of China Medical University, Shenyang, Liaoning, China